CLINICAL TRIAL: NCT07374458
Title: Effects of Esketamine and Bilateral Lower Limb Elevation on Hemodynamic Stability During Induction of General Anesthesia in Elderly Patients Undergoing Thoracic Surgery: A Factorial Design Study
Brief Title: Effects of Esketamine and Bilateral Lower Limb Elevation on Hemodynamic Stability During Induction of General Anesthesia in Elderly Patients Undergoing Thoracic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, XiaoLiang Wang, Principal Investigator, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: KY20251118-09
Record Dates: First submitted 2025-12-14; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Post Induction Hypotension
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Esketamine + Leg Elevation;Esketamine + Supine;Placebo + Leg Elevation;Placebo + Supine (Control) (Experimental): Esketamine + Bilateral Lower Limb Elevation:Participants received intravenous esketamine at a dose of 0.2 mg/kg, administered one minute before anesthesia induction. Bilateral Lower Limb Elevation Participants underwent bilateral lower limb elevation to 45°, initiated one minute before anesthesia induction.
  Esketamine + Supine Position:Participants received intravenous esketamine at a dose of 0.2 mg/kg, administered one minute before anesthesia induction.
  Placebo + Bilateral Lower Limb Elevation:Participants underwent bilateral lower limb elevation to 45°, initiated one minute before anesthesia induction.
  No Intervention: Placebo + Supine Position
  Interventions: Drug: Esketamine; Behavioral: Bilateral Lower Limb Elevation
- Esketamine + Supine Position (Experimental)
  Interventions: Drug: Esketamine
- Placebo + Bilateral Lower Limb Elevation (Experimental)
  Interventions: Behavioral: Bilateral Lower Limb Elevation
- Placebo + Supine Position (No Intervention)

INTERVENTIONS:
Drug: Esketamine — Participants received intravenous esketamine at a dose of 0.2 mg/kg, administered one minute before anesthesia induction.
  Arms: Esketamine + Leg Elevation;Esketamine + Supine;Placebo + Leg Elevation;Placebo + Supine (Control); Esketamine + Supine Position
Behavioral: Bilateral Lower Limb Elevation — Participants underwent bilateral lower limb elevation to 45°, initiated one minute before anesthesia induction.
  Arms: Esketamine + Leg Elevation;Esketamine + Supine;Placebo + Leg Elevation;Placebo + Supine (Control); Placebo + Bilateral Lower Limb Elevation

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) is widely used in thoracic surgery due to small incisions, low stress response, and high patient tolerance. Compared with open thoracotomy, VATS has fewer complications, shorter hospital stays, and better postoperative quality of life. Despite being minimally invasive, VATS can cause severe postoperative pain via pleural/lung parenchyma damage, intercostal nerve traction, and chest tube stimulation. This pain impairs patient mobility (e.g., turning over, getting out of bed), increasing risks of atelectasis and pulmonary infections. Approximately 78% of patients experience moderate-to-severe postoperative pain, and 50% receive inadequate analgesia [3]. Effective postoperative pain management is critical for recovery and reducing pulmonary infections. In recent years, combined general anesthesia with regional nerve blocks has been recommended to enhance postoperative comfort and accelerate recovery, as regional blocks alleviate pain and reduce general anesthetic dosage. Thoracic paravertebral block (TPVB), an effective regional anesthesia technique, is commonly used for postoperative analgesia in VATS.

TPVB involves injecting local anesthetics near thoracic spinal nerves exiting the intervertebral foramen, blocking ipsilateral somatic and sympathetic nerves. It is mainly used for analgesia after rib fractures, breast surgery, and thoracic surgeries (open or VATS). However, preoperative TPVB blocks both thoracic nerves and sympathetic nerves. Sympathetic inhibition reduces myocardial contractility, heart rate, and peripheral vascular resistance. Additionally, rapid administration of multiple drugs during general anesthesia induction further increases hypotension risk.

Esketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist, has stronger sedative/analgesic effects and fewer adverse events than ketamine. Studies show sub-anesthetic doses (0.15-0.3 mg/kg) reduce induction hypotension, opioid-induced cough, and other adverse events via sympathetic stimulation, analgesia, and NMDA receptor antagonism.

The passive leg raising (PLR) test assesses fluid responsiveness in acute circulatory failure by shifting ~300 mL of venous blood from lower limbs to the right heart. Its hemodynamic effects are reversible, avoiding fluid overload. Based on this, lower limb elevation during anesthesia induction rapidly and transiently increases venous return, reducing hypotension. Bilateral elevation enhances venous return, increases cardiac preload, improves cardiac output, and stabilizes blood pressure.

General anesthesia induction is a period of frequent hemodynamic fluctuations. Elderly patients, often with comorbidities and reduced physiological reserve, are more susceptible to induction-related hemodynamic disturbances (40% incidence). Sustained/severe hypotension causes inadequate organ perfusion/ischemia, increasing postoperative complications (myocardial injury, ischemic stroke, acute kidney injury). Preventing post-induction hypotension in the elderly is clinically valuable. Opioids, propofol, and muscle relaxants induce hypotension via arterial dilation and reduced peripheral resistance. TPVB-induced sympathetic block further increases hypotension risk. This study hypothesizes that esketamine administration or lower limb elevation during induction reduces hypotension incidence in elderly VATS patients with TPVB.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is now widely used in thoracic surgery due to its small incisions, low stress response, and high patient tolerance Compared to open thoracotomy, VATS is associated with fewer complications, shorter hospital stays, and better postoperative quality of life . Although VATS is a minimally invasive procedure, damage to the pleura and lung parenchyma, traction on the intercostal nerves, and stimulation from chest tubes can still cause severe postoperative pain. This pain affects patient mobility, such as turning over and getting out of bed, potentially leading to complications like atelectasis and pulmonary infections. Approximately 78% of patients experience moderate to severe pain after surgery, and 50% do not receive adequate analgesia [3]. Effective postoperative pain management is crucial for patient recovery and reducing pulmonary infections. To further ensure postoperative comfort and accelerate recovery, the combined use of general anesthesia with regional nerve blocks has been recommended in recent years. Regional blocks can not only effectively alleviate postoperative pain but also help reduce the dosage of general anesthetics, promoting faster patient recovery. Thoracic paravertebral block (TPVB), as an effective regional anesthesia technique, is often used to manage postoperative pain after VATS .

TPVB involves injecting local anesthetics near the thoracic spinal nerves as they exit the intervertebral foramen, blocking the ipsilateral somatic and sympathetic nerves. It is primarily used for analgesia following rib fractures, breast surgery, and open or video-assisted thoracic surgery. However, performing TPVB before surgery blocks both the thoracic nerves and the exposed sympathetic nerves. When sympathetic nerves are inhibited, myocardial contractility and heart rate decrease, while peripheral vascular resistance drops. Furthermore, the rapid administration of multiple drugs during general anesthesia induction can increase the incidence of hypotension during this period .

Esketamine is an N-methyl-D-aspartate (NMDA) receptor antagonist with stronger sedative and analgesic effects and fewer adverse events compared to ketamine. Some studies have shown that sub-anesthetic doses of esketamine (typically 0.15-0.3 mg/kg) can reduce the incidence of adverse events, such as induction hypotension and opioid-induced cough, through its sympathetic stimulatory, analgesic, and NMDA receptor antagonistic effects.

In cases of acute circulatory failure, the passive leg raising (PLR) test is used to assess whether cardiac output increases with volume expansion. By shifting approximately 300 mL of venous blood from the lower limbs to the right heart, PLR serves as a test of fluid responsiveness. Its hemodynamic effects can be quickly reversed by changing position, thus avoiding the risk of fluid overload. Based on this principle, elevating the patient's lower limbs during anesthesia induction can rapidly and transiently increase venous return to the heart, thereby reducing the occurrence of induction hypotension. Elevating both lower limbs enhances venous return from the legs, increasing preload to the heart, improving cardiac output, and helping to maintain stable blood pressure to some extent.

The induction period of general anesthesia is a phase of frequent hemodynamic changes. Elderly patients, often with multiple comorbidities and reduced physiological reserve, are more susceptible to hemodynamic disturbances caused by induction drugs. Studies indicate that approximately 40% of elderly patients experience hemodynamic alterations during induction . Sustained or severe hypotension may lead to inadequate organ perfusion and ischemia, potentially increasing the risk of postoperative complications such as myocardial injury, ischemic stroke, and acute kidney injury . Therefore, preventing hypotension after induction in elderly patients holds significant clinical value for reducing postoperative complications. The administration of opioids, propofol, and muscle relaxants during general anesthesia induction can cause hypotension due to arterial dilation and reduced peripheral vascular resistance. Since TPVB blocks sympathetic nerves, it may make patients more prone to hypotension during induction. This study hypothesizes that using esketamine or elevating the lower limbs during induction can reduce the incidence of hypotension in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-80 years old
* American Society of Anesthesiologists (ASA) physical status classification Ⅰ-Ⅲ
* Scheduled for elective thoracoscopic surgery under general anesthesia
* Informed consent: All patients or their family members voluntarily agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* Allergy to the drugs used in this study
* Severe cardio-cerebro-pulmonary diseases (including myocardial infarction, heart failure, cerebral hemorrhage, stroke, respiratory failure)
* Severe hepatic or renal diseases (Child-Pugh class C, or requiring renal replacement therapy)
* Severe neurological diseases (including Parkinson's disease, Alzheimer's disease)
* History of poorly controlled hypertension, or systolic blood pressure > 180 mmHg or mean arterial pressure (MAP) < 70 mmHg before anesthesia induction
* Increased intracranial pressure, glaucoma, penetrating ocular trauma, or moderate to severe pulmonary arterial hypertension
* Spinal diseases (deformity or trauma), history of spinal surgery, abnormal skin sensation of the chest and back, infection at the puncture site, or abnormal coagulation function
* Abdominal hypertension or lower extremity deep vein thrombosis
* Emergency surgery
* Body mass index (BMI) ≥ 35 kg/m²

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypotension | From the start of anesthesia induction to 5 minutes after induction

SECONDARY OUTCOMES:
Incidence of Severe Hypotension | From the start of anesthesia induction to 5 minutes after induction
Postoperative Esketamine-Related Adverse Effects | Within 24 hours after surgery
  Incidence of headache, dizziness, nightmares, and mood disturbances following esketamine administration.
Postoperative Sleep Quality | Within 24 hours after surgery
  Sleep quality assessed by the Richards Campbell Sleep Questionnaire (RCSQ),"Sleep quality was assessed using the Richards-Campbell Sleep Questionnaire (RCSQ), which ranges from 0 to 100, where higher scores represent better sleep quality."
Use of Vasoactive Medications During Anesthesia Induction | From the start of anesthesia induction to 5 minutes after induction
  Record whether vasoactive medications were administered during anesthesia induction.
Stroke Volume During Anesthesia Induction | From the start of anesthesia induction to 5 minutes after induction
  Stroke volume measured during anesthesia induction
Cardiac Index During Anesthesia Induction | From the start of anesthesia induction to 5 minutes after induction
  Cardiac index measured during anesthesia induction.
Oxycodone Consumption Within 24 Hours After Surgery | Within 24 hours after surgery
  Total oxycodone consumption recorded from the postoperative analgesia pump.
Time to First Analgesia Pump Activation | Within 24 hours after surgery
  Time from arrival in the recovery area to the first activation of the postoperative analgesia pump.
Number of Effective Analgesia Pump Activations | Within 24 hours after surgery
  Number of effective activations of the postoperative analgesia pump.
Postoperative Recovery Quality | 24 hours after surgery
  Quality of postoperative recovery assessed using the Quality of Recovery-15 (QoR-15) questionnaire, a validated patient-reported outcome measure. The total score ranges from 0 to 150, with higher scores indicating better quality of recovery.
Postoperative Pain Scores | 4 and 24 hours after surgery
  Postoperative pain intensity assessed using the Visual Analog Scale (VAS), a validated pain assessment tool ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Pain scores were assessed at rest and during movement (coughing).
Intraoperative Cough | From the start of anesthesia induction to 5 minutes after induction
Postoperative Complications | From induction to 24 hours after surgery
  Record cough during induction, and postoperative nausea, vomiting, and delirium incidence
Patient Satisfaction | Within 72 hours after surgery
  Patient satisfaction with perioperative care assessed using a 5-point Likert scale, ranging from 1 (very dissatisfied) to 5 (very satisfied).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR, Analytic Code